CLINICAL TRIAL: NCT02132572
Title: Retrospective Multi-centre, Post-marketing Study to Evaluate the Incidence and Aetiology of Reoperations With Allergan Natrelle® Breast Implants in Primary Augmentation (RANBI)
Brief Title: Retrospective Study of Incidence and Etiology of Reoperation After Primary Augmentation With Natrelle® Breast Implants
Acronym: RANBI
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF-AGN-MED-BRE-003
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Natrelle BIOCELL™ Textured 410 Implant: Previously received a Natrelle BIOCELL™ textured 410 implant for primary breast augmentation.
  Interventions: Device: BIOCELL™ Textured 410 Implant

INTERVENTIONS:
Device: BIOCELL™ Textured 410 Implant — Previously received a Natrelle BIOCELL™ textured 410 implant for primary breast augmentation.

SUMMARY:
Retrospective multi-center, post-marketing study to evaluate the incidence and etiology of reoperations with Allergan Natrelle® Breast Implants in primary augmentation (RANBI)

ELIGIBILITY:
Inclusion Criteria:

* Primary breast augmentation (either bilateral or unilateral) operated on by the investigating surgeon with an infra-mammary approach 410 cohesive BIOCELL™ textured device (Truform 2 & 3 only) has been implanted
* Primary breast augmentation 3 to 10 years prior to data collection
* Submuscular/dual plane or subglandular implant placement

Exclusion Criteria:

* Breast augmentation for Poland Syndrome or amastia
* Breast reconstruction following mastectomy
* Revision or secondary breast reconstruction
* Non 410 device at initial breast augmentation
* Women subsequently diagnosed with fibrocystic disease considered to be pre-malignant
* Procedures of the breast not related to the primary breast augmentation (e.g. excision of skin lesions)
* Axillary or peri-areolar approach
* Glandular mastopexy augmentation (skin excision only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have undergone a primary breast augmentation for aesthetic reasons with a Natrelle BIOCELL™ textured 410 cohesive implant
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (5):
- Bordeaux, France
- Düsseldorf, Germany
- Tel Aviv, Israel
- Madrid, Spain
- East Grinstead, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natrelle BIOCELL™ Textured 410 Implant
Started | 201
Completed | 201
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Natrelle BIOCELL™ Textured 410 Implant
Number analyzed (Participants) | 201
Age, Customized [Number; unit: Participants]
  17 to 30 years | 67
  31 to 40 years | 74
  41 to 50 years | 36
  51 to 60 years | 18
  61 to 70 years | 3
  Missing age data | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With First Reoperation Following Use of a BIOCELL™ Textured 410 Implant
Description: Data were retrospectively collected on the percentage of subjects who had a first reoperation following previous breast augmentation with a BIOCELL™ Textured 410 Implant.
Time Frame: 3 to 10 years
Population: Per Protocol: Subjects who underwent a primary breast augmentation with BIOCELL™ textured 410 cohesive breast implants 3 to 10 years prior to data collection
Measure: Number; unit: Percentage of Subjects
Arm/Group | Natrelle BIOCELL™ Textured 410 Implant
Number analyzed (Participants) | 175
Percentage of Subjects | 28

ADVERSE EVENTS:
Description: The Safety Population included all subject who underwent a primary breast augmentation with BIOCELL™ textured 410 cohesive breast implants for aesthetic reasons. The Safety Population was used to assess adverse events and serious adverse events.
Arm/Group | Natrelle BIOCELL™ Textured 410 Implant
Serious Adverse Events (participants affected / at risk) | 30/201
Other Adverse Events (participants affected / at risk) | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natrelle BIOCELL™ Textured 410 Implant (N=201)
Device Breakage (General disorders) | 7
Device Dislocation (General disorders) | 8
Capsular Contracture Associated with Breast Implant (General disorders) | 7
Device Optical Issue (General disorders) | 6
Device Damage (General disorders) | 2
Device Deployment Issue (General disorders) | 1
Device Expulsion (General disorders) | 1
Impaired Healing (General disorders) | 1
Implant Site Reaction (General disorders) | 2
Nipple Disorder (Reproductive system and breast disorders) | 1
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast Pain (Reproductive system and breast disorders) | 1
Device Issue (General disorders) | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 5
Scar Excision (Surgical and medical procedures) | 1
Seroma (Injury, poisoning and procedural complications) | 4
Surgery (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.